CLINICAL TRIAL: NCT04294823
Title: Sensitivity and Specificity of the Modified Helicobacter Test INFAI Using New Test Meal With Urea Breath Test in Helicobacter Pylori Positive and Negative Patients With Dyspepsia and GERD Taking Proton Pump Inhibitors
Brief Title: Sensitivity and Specificity of the Modified Helicobacter Test INFAI
Status: Withdrawn | Type: Observational
Why Stopped: Administrative delays were too long
Sponsor: International Pharmaceutical Consultancy (Other)
Responsible Party: Sponsor
Other Study IDs: HPT30/J/17
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Dyspepsia; GERD
MeSH Terms: conditions — Dyspepsia; Gastroesophageal Reflux | interventions — Endoscopy; Gastroscopy; Esomeprazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FRANCE - CHU creteil: An internal physical examination including vital signs measurements and a 13C-UBT with the standard test meal (Helicobacter Test INFAI) will be performed. Patients with a positive UBT will undergo upper endoscopy. All biopsy samples will be analysed in the local laboratory of the centre. Patients with a negative UBT will undergo also upper endoscopy. Endoscopic procedures and subsequent investigations will be identical in patients with a positive and with a negative UBT. H. pylori positive and negative patients will perform the 13 C-UBT breath tests with new test meal on Day 30. The study will be conducted in outpatients. Starting on Day 1, H. pylori positive and negative patients will take Nexium mups 40 mg orally once daily, 30 min before breakfast. Patients will return to the hospital/medical practice for UBT breath tests with new test meal on Day 30. Patients will be followed-up for 7 days after discontinuation of PPI treatment.
  Interventions: Diagnostic Test: Helicobacter Pylori Diagnostic; Device: Vital signs measurments; Diagnostic Test: endoscopy; Drug: Nexium Pill

INTERVENTIONS:
Diagnostic Test: Helicobacter Pylori Diagnostic — Helicobacter Test INFAI with standard test Meal (1g citric acid as test meal and 75 mg C^13 urea)
  + The C^13 UBT with the new test (REFEX). All patients will take Nexium mups (40 mg) orally once daily 30 min before breakfast from day 1 to 28.
  Other Names: Helicobacter test INFAI
Device: Vital signs measurments — No description;
Diagnostic Test: endoscopy — Upper endoscopy where 6 biopsy samples will be obtained . Two biopsies will be taken from antrum and corpus for histology. The biopsies will be stained with Haematoxylin & Eosin and Giemsa stains, and gastritis wilt be scored using the Updated Sydney System 12,13 Two biopsies will be taken from antrum and corpus for rapid urease test (RUT) and two biopsies will be taken from antrum and corpus for culture. All biopsy samples will be analysed in the local laboratory of the centre.
  Other Names: Upper endoscopy
Drug: Nexium Pill — patients will take Nexium mups 40 mg orally once daily, 30 min before breakfast Nexium mups 40 mg will be discontinued after Day 28.

SUMMARY:
Study to confirm the sensitivity of the C^13-UBT using the new test meal for H. Pylori in patients with dyspepsia and GERD taking PPI

Secondary objectives : to compare the sensitivity and specificity of the C^13-UBT using the new test meal and standard test meal for H.Pylori in patients with dyspepsia and GERD taking PPI.

to complete the results of the Helicbacter test INFAI using new test meal for H.Pylori in patients with dyspepsia and GERD taking PPI with :

* Histology score for H.Pylori in antrum an corpus using the updated Sydney System
* Sex,
* Age,
* Body Mass Index (BMI)

DETAILED DESCRIPTION:
Helicobacter pylori (H. pylori) infection can be diagnosed by invasive (i.e., endoscopy and biopsy) and non-invasive techniques . The most accurate non-invasive tests for diagnosing active H. pylori are the 13C-urea breath test and the stool antigen test3 Several guidelines for the management of dyspeptic patients in primary care settings recommend the use of non-invasive tests for H. pylori in the initial management of dyspeptic patients (test and treat strategy)3 . This strategy has been tested in a number of clinical settings and has been shown to be effective from both a clinical and a cost perspective The urea breath test (UBT) and the stool antigen test are very sensitive and specific except in patients taking proton pump inhibitors (PPI) 678 In patients taking PPI, a positive test remains reliable for the detection of H. pylori but the number of false negative tests rises dramatically reducing the sensitivity of these tests. PPI are widely available and are over-thecounter agents in some countries (e.g. USA, Sweden). Clinicians are frequently confronted with making a diagnosis of H. pylori infection in patients who may knowingly or unknowingly be taking PPI. Currently available breath and stool tests are reliable 12 - 14 days after discontinuation of the PPI. This results in the cost and inconvenience of another visit and the possibility of symptoms in some patients when the PPI is withdrawn.

Although the exact mechanism by which acid inhibition causes a false negative reaction is unclear, some studies have suggested that acidification of the stomach may reverse the abnormality Results have been inconsistent, however, and how to acidify the stomach and to what extent this should be done is unclear. Standardised test meals are routinely administered with the breath test substrate.

The aim of this study is to assess the sensitivity and specificity of the 13C-urea breath test administered with the new test meal in patients with dyspepsia and GERD taking PPI.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients of at least 18 years of age.
* All acid-related disorders requiring long-term PPI treatment including functional dyspepsia according Rome IV classification.
* Positive or negative standard 13C-UBT at screening.
* Diagnosis of H. pylori infection confirmed or excluded by combination of culture , histology and rapid** urease test (PyloriTek@, Serim Research Corp., Elkhart, IN, USA) on samples obtained by endoscopy:
* True positive if culture positive and/or positive histology in combination with positive urease test.
* True negative if culture is negative and if histology and/or urease test is negative. True negative if culture not evaluable and both histology and urease test are negative.
* Culture will be based on biopsies from antrum and corpus. Two biopsies will be taken from antrum and corpus for histology. Rapid urease test will be performed on the samples of antrum and corpus. Written informed consent of the patient.

Exclusion Criteria:

* Previous H. pylori eradication therapy.
* Intake of PPI off 14 days, 1-12 receptor antagonists 1 day, NSAlDs, antibiotics, antisecretory drugs, bismuth compounds, or sucralfate in the 4 weeks prior to enrolment.
* Manifest coagulopathy or any other disorder according to which endoscopy and/or biopsies are contraindicated.
* Participation in a clinical trial with another not approved drug within 30 days before entering the study and/or previous participation in this study.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A minimum of 57 H. pylori positive patients and a minimum of 57 H. pylori negative patients fulfilling all inclusion criteria and none of the exclusion criteria will be included
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-11 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
13C-breath test | 1 month
  In every breath sample the 13C02 / total C02 ratio will be determined at baseline and at 30 min after ingestion of the urea-BC solution.
  The delta over baseline (DOB) or Aö-value [0/00] will be calculated from the difference of the 13C02 / total C02 ratio 30 min after intake of the BC solution and at baseline. urea- The test for the standard test meal is positive if DOB or the A6-vaIue is greater than 4 0/00.
  The test for the new test meal is positive if DOB or the A6-vaiue is greater than 2.5 0/00. Coefficients of correlation between DOB and the histology score for H. pylori in antrum and corpus using the Updated Sydney System, sex, age and BMI.

CONTACTS AND LOCATIONS:
Locations (1):
- CHI de créteil, Créteil, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No